CLINICAL TRIAL: NCT06863675
Title: Highly Aspherical Lenslet (HAL) and Binocular Vision (BV) Disorders [HALT X(T) Study]
Acronym: HALT XT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Bryan Sim XR, Consultant, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SingaporeNEC_HALTXT
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Myopia; Strabismus
Keywords: Myopia; Strabismus; HALT; Stellest; Myopia Control
MeSH Terms: conditions — Myopia; Strabismus

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial (RCT)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HALT lenses for children with strabismus (Active Comparator): Stellest lenses for children with strabismus
  Interventions: Device: HAL lenses for children with strabismus
- SVL for children with strabismus (Placebo Comparator): SVL for children with strabismus
  Interventions: Device: SVL for children with strabismus

INTERVENTIONS:
Device: HAL lenses for children with strabismus — It has been shown that peripheral segmented defocus spectacles can slow myopia progression. The Essilor® Stellest™ lens has been designed with an exclusive and pioneering technology called HALT (Highly Aspherical Lenslet Target). The HALT technology is made of a constellation of 1,021 invisible lenslets. This constellation creates a signal in front of the retina that acts as a shield against eye elongation and, therefore, myopia progression. Studies suggest that children are tolerable against these glasses, and the lenses can slow down myopia progression by 67% on average, compared to single vision lenses, when worn 12 hours a day. It can be considered as one of the best available myopia control spectacle lens designs, being superior to progressive addition and bifocal lenses.
  Arms: HALT lenses for children with strabismus
Device: SVL for children with strabismus — SVL for children with strabismus
  Other Names: Single Vision Lenses
  Arms: SVL for children with strabismus

SUMMARY:
Assess the effect and changes of eye misalignment (strabismus) with myopia control glasses Assess the efficacy of myopia control glasses on childhood myopia progression in children with strabismus due to the uncertainty clinicians face when prescribing myopia control glasses to these strabismic children

DETAILED DESCRIPTION:
Studies have been done to show that spectacles, atropine eye drops, and outdoor activities have some efficacy in slowing myopia progression in children, however most of such studies exclude children with significant eye conditions such as strabismus or nystagmus to isolate the effects of myopia control treatment. In this study, we would like to investigate whether these specialized glasses can effectively slow down the progression of myopia in children with strabismus. Since strabismus can affect visual development, this study would also be able to assess the effect and changes of eye misalignment (strabismus) with myopia control glasses. The study also aims to assess the efficacy of myopia control glasses on childhood myopia progression in children with strabismus due to the uncertainty clinicians face when prescribing myopia control glasses to these strabismic children.

ELIGIBILITY:
Inclusion Criteria:

Age 5-12 years old Myopia of between -1D and -6D in at least 1 eye Progression of at least 0.5D within the last year Astigmatism less than 2.5D Exotropia Exophoria: horizontal deviation <40PD Esotropia (good control), Esophoria: horizontal deviation <40PD Any vertical strabismus: Vertical deviation <10 PD Intermittent exotropia (good, moderate, poor) Horizontal deviation ≥15 PD, vertical deviation ≤5 PD (?)

Exclusion Criteria:

VA poorer than logMAR 0.2 (6/9.5) in either eye Any other ocular condition (e.g. lens opacity, glaucoma) other than myopia, strabismus or nystagmus) Any medical/neurological condition which would interfere with subjects ability to co-operate with tests and attend follow-up appointments.

Plans of surgery for strabismus or nystagmus in the next year Constant XT). Past use of any other from of myopia control treatment (eg. atropine or myopia control glasses or contact lenses) within the last year.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of HAL lenses in childhood myopia control in children with strabismus and nystagmus | 2 years
  a. Efficacy in each eye - i. Primary outcome: change in AL in first vs second 6m ii. Secondary outcome: change in cycloplegic SE & OCT choroidal thickness b. Alternative analysis: Difference between preferred/non-preferred eye, better-worse squint (size and control at baseline and 6m).

SECONDARY OUTCOMES:
To assess the effect on strabismus (subjectively and functionally) over first vs second 6m | 2 years
  Primary measure: Change in squint size and control as measured by Newcastle control score (NCS)

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Inclusion exclusion criteria Age Myopia progression Axial length
Supporting Information: Study Protocol, ICF, CSR
Time Frame: June 2025 to June 2028
Access Criteria: PI Co-PI Study members